CLINICAL TRIAL: NCT02905968
Title: The Safety and Effect of Transanual Tube Placement in Low Anterior Resection (LAR) for Rectal Cancer to Prevent Anastomotic Leak: Randomized Control Trial Study
Brief Title: Transanual Tube Placement in Low Anterior Resection (LAR) for Rectal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTPLAR
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Rectal Cancer
Keywords: Anastomotic leak; Low rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TTPLAR (Experimental): Transanual tube placement after anastomosis in low anterior resection for rectal cancer.
  Interventions: Device: transanual tube placement
- NORLAR (No Intervention): Tranditional low anterior resection without transanual tube placement or ileostomy.

INTERVENTIONS:
Device: transanual tube placement — Transanual tube placement after anastomosis in low anterior resection for rectal cancer.
  Arms: TTPLAR

SUMMARY:
The purpose of this study is to evaluate the effectiveness of transanual tube placement in low anterior resection (LAR) for rectal cancer in preventing anastomotic leakage.

DETAILED DESCRIPTION:
Transanual tube placement after anastomosis in low anterior resection for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Primary tumor has undergone histologically confirmed rectal adenocarcinoma; Low rectal cancer was defined by the presence of the inferior pole of the tumor below the peritoneal reflection (in 11 cm from the anal margin).
3. Together with clinical or radiological evidence of Stage II (T3-4, N0, M0) or Stage III (T1-4, N1-2, M0) disease (according to the 2010 revision of the International Union Against Cancer primary tumor, regional nodes, metastasis (TNM) staging system).
4. Performance status (ECOG) 0~1
5. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; hemoglobin (Hb) ≥9g/dl (within 1 week prior to randomization)
6. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either primary tumor, regional nodes, metastasis (AST) or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
7. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Body mass index (BMI) more than 30 kg/m2.
2. Serious pre-operative comorbidity, including cardiovascular disease (coronary arteriosclerosis, arrhythmia, heart failure), pulmonary dysfunction (lung emphysema, obstructive lung disease), liver insufficiency (Child-Pugh B or C), renal insufficiency (serum creatinine >2.0 mg/dl), and arterial circulation disturbance (occlusion of arterial vessels of limb in patient's history.
3. History of accepting abdominal surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak rate | 30 days post operatively
  Anastomotic leak is a common and serious complication after low anterior, resection, and often leads to re-operation.

SECONDARY OUTCOMES:
Time Frame: Reoperation rate after anastomotic leak | 30 days post operatively
  Anastomotic leak is a common and serious complication after low anterior, resection, and often leads to excrement peritonitis, and re-operation as colostomy

CONTACTS AND LOCATIONS:
Overall Officials: Tuo Yi, MD, Principal Investigator — Fudan University
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China